CLINICAL TRIAL: NCT05704205
Title: The UPDATE Trial (Uvb Phototherapy in Dermatology for ATopic Eczema): A Multicenter Randomized Controlled Trial of Narrowband UVB Versus Optimized Topical Therapy in Patients With Atopic Eczema
Brief Title: The UPDATE Trial (Uvb Phototherapy in Dermatology for ATopic Eczema)
Acronym: UPDATE
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other)
Collaborators: ZonMw: The Netherlands Organisation for Health Research and Development (Other)
Responsible Party: Principal Investigator, Prof. Dr. Phyllis I. Spuls, Principal Investigator, Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NL81882.018.22
Record Dates: First submitted 2022-12-08; First posted 2023-01-30 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2026-01

CONDITIONS: Atopic Dermatitis Eczema; Atopic Dermatitis
Keywords: atopic eczema; atopic dermatitis; NB-UVB; phototherapy; optimal topical therapy
MeSH Terms: conditions — Dermatitis, Atopic

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial
Who Masked: Outcomes Assessor
Masking Description: Single blinded
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- NB-UVB+OTT (Experimental): 8-16 weeks of NB-UVB phototherapy combined with (a minimum of) 3 months of optimal topical therapy
  Interventions: Device: NB-UVB phototherapy; Combination Product: Optimal topical therapy
- Optimal topical therapy (OTT) (Active Comparator): (a minimum of) 3 months of optimal topical therapy
  Interventions: Combination Product: Optimal topical therapy

INTERVENTIONS:
Device: NB-UVB phototherapy — Narrowband ultraviolet B irradiation 3 times a week
  Other Names: Narrowband ultraviolet B phototherapy
  Arms: NB-UVB+OTT
Combination Product: Optimal topical therapy — A combination of detailed instructions about the disease and treatments by trained nurses, bathing and washing advices, adequate emollients use, avoidance of triggers (including possible and proven contact allergens), fingertip unit explanation for active topical therapy, and personalized topical therapy with different potency topical steroids, calcineurin inhibitors and tar ointments
  Other Names: OTT; Optimal local therapy

SUMMARY:
The goal of this randomized controlled trial is to study the (cost)effectiveness of NB-UVB phototherapy in patients with atopic eczema/atopic dermatitis.

Half of the participants will undergo a course of NB-UVB phototherapy of 8-16 weeks and apply optimal topical therapy (OTT) for a minimum of 3 months. Researchers will compare the outcomes of this group with the other half of participants that apply OTT only.

DETAILED DESCRIPTION:
Atopic eczema (AE) is a chronic fluctuating dermatological disease characterized by a pruritic inflammation of the skin. The condition poses a high global (financial) burden. One of the therapeutic options of AE is phototherapy, with narrowband UVB (NB-UVB) being the most common. The evidence of the (cost-)effectiveness of NB-UVB, however, is scarce and of low quality.

The objective of this pragmatic multicenter single blinded randomized controlled trial is comparing the effectiveness and cost-effectiveness of narrowband ultraviolet B with optimal topical therapy (NB-UVB+OTT) versus OTT at 3 months in adult patients with insufficient control of their AE with standard topical treatment, for whom dermatologist and patient jointly believe that NB-UVB or OTT is needed.

Participants that are randomized into the NB-UVB+OTT group will receive an NB-UVB course (at home or at the outpatient clinic) for at least 8 and up to 16 weeks, combined with OTT for at least 3 months. Participants in the control group (OTT group) will apply OTT for at least 3 months. Visits will occur at baseline and 1-3-6-9-12 months after start. At baseline, patient information is collected including an evaluation of medical history and a physical examination to assess Fitzpatrick skin type and physician-reported clinical signs. During each visit patients are asked to fill out questionnaires. Risks are expected to be as in daily practice.

Primary study parameters/outcome of the study is the percentage of patients with EASI50 (a decrease of the Eczema Area and Severity Index of 50%) at 3 month follow-up. Secondary study parameters/outcome of the study include delta EASI, physician-reported clinical signs, patient-reported symptoms, quality of life, long-term control, cost-effectiveness, side effects at 1-3-6-9-12 months, quantity and potency topical steroid usage, time to starting systemic therapy, patient satisfaction with received treatment, percentage of patients reaching Treatment Target goals and percentage of drop-outs with reasons at 3-6-9-12 months.

ELIGIBILITY:
Inclusion Criteria:

* Adult (≥18 years of age) patient meeting the UK working party criteria for atopic eczema;
* AE insufficiently controlled by standard topical care and therefore eligible for NB-UVB or OTT;
* Investigator Global Assessment (IGA, 0-4) of ≥ 2 (moderate disease);
* Eczema Area and Severity Index (EASI) of ≥ 7 (moderate disease);
* Understood and voluntarily signed and dated an informed consent form prior to any study-related procedure or has a legal representative who has, and is willing to comply with the study's requirements.

Exclusion Criteria:

* Contra-indication for NB-UVB;

  * Genetic defects associated with photosensitivity or skin cancer;
  * Heavily photo-damaged skin;
  * History of multiple (>1) skin malignancies;
  * Use of systemic immunosuppressants/immunomodulators;
  * Use of medication associated with photosensitivity;
* Patient is already on systemic AE therapy;
* Patient is already on OTT in the past 2 months;
* NB-UVB or any systemic therapy in the past 9 months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 316 (Estimated)
Dates: Start 2023-02-22 (Actual); Primary Completion 2026-01-16 (Actual); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Percentage of patients that reach EASI50 | 3 months
  Percentage of patients that reach a 50% reduction of the EASI (Eczema Area and Severity Index) at 3 month follow-up

SECONDARY OUTCOMES:
Delta EASI | 3 months
  Change in EASI (Eczema Area and Severity Index) at 3 month follow up
Cost-effectiveness | 1 year
  Questionnaire-based calculation of medical consumption- and productivity costs in both arms
Patient reported outcomes | 1 year
  Questionnaire-based review of quality of life, patient satisfaction
Time to start systemic therapy | 1 year
  The time to start of systemic AE treatment in both arms
Quantity of topical steroid usage | 1 year
  The amount of used topical corticosteroids in both groups
Potency of topical steroid usage | 1 year
  The potency (I-IV) of used topical corticosteroids in both groups

CONTACTS AND LOCATIONS:
Overall Officials: Louise AA Gerbens, MD PhD, Principal Investigator — Amsterdam University Medical Centers
Locations (16):
- Netherlands (16):
  - Flevoziekenhuis, Almere Stad, Flevoland
  - Jeroen Bosch Ziekenhuis, 's-Hertogenbosch, North Brabant
  - Centrum Oosterwal, Alkmaar, North Holland
  - OLVG, Amsterdam, North Holland
  - Amsterdam Universitair Medische Centra, Amsterdam, North Holland
  - Huid Medisch Centrum, Amsterdam, North Holland
  - Bergman Clinics, Haarlem, North Holland
  - Spaarne Gasthuis, Hoofddorp, North Holland
  - Dijklander Ziekenhuis, Purmerend, North Holland
  - Isala Klinieken, Zwolle, Overijssel
  - Medisch Centrum Leeuwarden, Leeuwarden, Provincie Friesland
  - Reinier de Graaf Gasthuis, Delft, South Holland
  - Leids Universitair Medisch Centrum, Leiden, South Holland
  - Alrijne Ziekenhuis, Leiderdorp, South Holland
  - Erasmus Medisch Centrum, Rotterdam, South Holland
  - Meander Medisch Centrum, Amersfoort, Utrecht

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Knops E, Spuls P, Duijnhoven R, Dijkgraaf M, van Barreveld M, Arents B, van Enst A, Garritsen F, Merkus M, Middelkamp-Hup MA, Musters A, Bosma A, Hyseni A, Dijkstra J, Hijnen DJ, Gerbens L. The UPDATE trial (UVB Phototherapy in Dermatology for ATopic Eczema): study protocol for a randomized controlled trial of narrowband UVB with optimal topical therapy versus optimal topical therapy in patients with atopic eczema. Trials. 2024 Jul 16;25(1):482. doi: 10.1186/s13063-024-08334-z. PMID 39014498